CLINICAL TRIAL: NCT00238693
Title: Transplant Registry: Patients Who May Require Transplantation and Those Who Have Undergone Transplantation of Liver, Kidney and/or Pancreas
Brief Title: Transplant Patient Registry of Liver, Kidney and/or Pancreas
Status: Completed | Type: Observational
Sponsor: Virginia Commonwealth University (Other)
Responsible Party: Sponsor
Other Study IDs: HM3127
Record Dates: First submitted 2005-10-11; First posted 2005-10-13 (Estimated); Last update posted 2018-09-25 (Actual); Status verified 2018-09

CONDITIONS: End Stage Renal Disease; End Stage Liver Disease
Keywords: transplant; transplantation of liver, kidney, pancreas
MeSH Terms: conditions — Kidney Failure, Chronic; End Stage Liver Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This is a registry of data collected from patient records, both of those who have a condition which may require transplantation and those who have undergone transplantation of the liver, kidney and/or pancreas.

DETAILED DESCRIPTION:
Honest Broker arrangement.

ELIGIBILITY:
Inclusion Criteria:

* Patients followed in the transplant clinic at Virginia Commonwealth University Health System

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients followed in the transplant clinic at Virginia Commonwealth University Health System
Sampling Method: Probability Sample
Enrollment: 13767 (Actual)
Dates: Start 2003-04; Primary Completion 2018-08-27 (Actual); Study Completion 2018-08-27 (Actual)

PRIMARY OUTCOMES:
Data collection and maintenance | Ongoing
  MAINTAIN A CURRENT, ACCURATE DATA BASE OF TRANSPLANT RECIPIENTS WITH REGARDS TO TRANSPLANT DATA AND OUTCOMES.

CONTACTS AND LOCATIONS:
Overall Officials: Adrian H Cotterell, MD, FACS, Principal Investigator — Virginia Commonwealth University Health System
Locations (1):
- Virginia Commonwealth University Health System, Richmond, Virginia, United States